CLINICAL TRIAL: NCT07358832
Title: Neuromodulation Through Multisensory Stimulation for Visual Field Deficits in the Subacute Stage of Disease
Acronym: MULTICAMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25C504
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Homonymous Hemianopsia; Stroke
MeSH Terms: conditions — Hemianopsia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal Occipital tDCS + audio-visual training (Experimental): Anodal tDCS on ipsilesional occipital cortex. Anode electrode placed on O1/O2 (10-20 EEG system) and reference electrode placed on the contralateral forehead. Stimulation delivered at 2mA during the first 30 minutes of the audio-visual training.
  Interventions: Device: tDCS; Behavioral: Audio-visual training
- Sham tDCS + audio-visual training (Sham Comparator): Same montage as for Experimental group. Stimulator is turned off after 30s of the audio-visual training.
  Interventions: Device: tDCS; Behavioral: Audio-visual training

INTERVENTIONS:
Device: tDCS — Anodal or sham tDCS (see "Arms") is applied during the execution of an audio-visual training.
Behavioral: Audio-visual training — 90 min/day x 10 days. Participants are seated in front of a 2 m × 2 m training board, at a distance of 1.2 m, in a dimly lit room. The board features 48 red light-emitting diodes (LED, diameter 1 cm, luminance 90 cd m2), distributed in six horizontal rows (eight lights per row). Forty-eight piezoelectric loudspeakers (0.4 W, 8Ω) are located above each light, producing a white-noise (80 dB, duration 100 ms).
  Spatio-temporally congruent, cross-modal, audio-visual stimuli are presented at one out of 48 possible positions on the board. Participants are instructed to look at the fixation point - at the center of the apparatus - and to move their eyes to detect the presence of the visual stimulus (duration=100 ms) by pressing right button of a wireless mouse.

SUMMARY:
Homonymous visual field defects (HVFDs) after acquired brain injuries affect daily life by impairing reading, navigation, and social activities, often impacting anxiety and depression. Spontaneous recovery is rare. Rehabilitation approaches include restorative treatments, which aim to expand the visual field through the stimulation of the so-called transition zone, and compensatory strategies, such as audio-visual training (AVT), which combines eye movement exercises with synchronized visual and auditory cues to train oculomotor scanning and overcome the visual field loss. Combining AVT with non-invasive brain stimulation, such as transcranial direct current stimulation (tDCS), may enhance recovery by promoting brain plasticity. Early evidence suggests that tDCS applied to the lesioned visual cortex during AVT can speed and stabilize improvements, potentially also restoring parts of the visual field. However, most studies on AVT have focused on chronic patients, whereas several clinical trials and international guidelines indicate that early treatment of HVFDs in the subacute phase can optimally exploit the window of maximal neural plasticity and prevent secondary degenerative processes, thereby maximizing visual recovery.

In the present randomized clinical trial, we assess the efficacy of a multisensory audio-visual training (AVT) combined with tDCS in patients with subacute HVFDs after stroke (<3 months post-lesion). Participants are randomly assigned to two groups: AVT combined with real anodal tDCS applied to the lesioned occipital cortex (Group 1), or AVT combined with sham tDCS (Group 2).

The AVT requires participants to orient their gaze toward spatio-temporally congruent, cross-modal audio-visual stimuli (starting from a central fixation) and press a button as quickly as possible upon detecting the visual target. All stimuli are presented on 2mx2m panel embedded with 40 LEDs and loudspeakers (Diana, Casati, Melzi, Marzoli, et al., 2024). The training will be administered for 90 minutes daily over 10 consecutive days.

All participants underwent a neuro-ophthalmological evaluation and neuropsychological assessment of visuospatial functions before the beginning of the training (t0), at the end of the training (t1), at 2 months (t2) and after 1 year (t3).

ELIGIBILITY:
Inclusion Criteria:

- Presence of subacute acquired brain injury (< 3 months) with HVFD according to Neurophthalmological evaluation

Exclusion Criteria:

* Presence of hemispatial neglect (indexed by pathological asymmetries on paper-and-pencil tests)
* Disorders of conjugated eye movements
* Other neurological disorders (e.g., dementia)
* Exclusion criteria for brain stimulation (i.e., epilepsy or family history of epilepsy; implanted electrodes, stimulators, pacemakers, infusion pumps, or any implanted metal device; pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Humphrey Visual Field perimetry | At baseline (at the beginning of the treatment), at the end of the treatment, at 2- and 12-month follow-ups
  Mean Deviation (MD) values of both eyes will be averaged and used for the analyses. Negative values will reflect a deviation from the expected performance in the participant's age group, hence a visual field defect.

SECONDARY OUTCOMES:
Change from baseline in Accuracy and reaction time on the EF Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 2- and 12-month follow-ups
  Computerized visual search task. Participants have to search for the target letter "F" surrounded by distractors "E"s. Accuracy: the proportion of correct responses (range 0-1). RTs: median search times (seconds) of correct responses.
Change from baseline in Accuracy and Reaction times on the Triangle Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 2- and 12-month follow-ups
  Computerized visual search task. Participants have to report the number of triangles (targets) surrounded by square distractors. Accuracy: the proportion of correct responses (range 0-1). RTs: median search times (seconds) of correct responses.
Change from baseline in Accuracy and RTs on the Visual Detection Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 2- and 12-month follow-ups
  Detection of visual stimuli presented on the same panel employed for the training. Accuracy (the proportion of detected stimuli; range 0-1) is calculated for both the sighted and the blind hemifields. RTs: median search times of the detected stimuli are calculated for both the sighted and the blind hemifields.
Change in retinal layers thickness assessed with Spectral Domain Optical Coherence Tomography | At baseline (at the beginning of the treatment), at 2- and 12-month follow-ups
  Non-invasive medical imaging technique that uses light waves to create high-resolution, cross-sectional pictures (tomograms) of retinal layers. We will assess the peripapillary retinal nerve fiber and the macular ganglion cell complex layers
Change in Visual Evoked Potential amplitude | At baseline (at the beginning of the treatment), at the end of the treatment and at 12-month follow-ups
  We will record with electroencephalography pattern reversal VEPs from monocular stimulation of each visual hemifield. We will analyzed the amplitude of P100 component.
Change from baseline in the functional scale assessing the impact of vision loss in everyday life activities | At baseline (at the beginning of the treatment), at the end of the treatment, at 12-month follow-ups
  We will use the 25-item National Eye Institute Visual Function Questionnaire. The total score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy